CLINICAL TRIAL: NCT06110299
Title: Room Air vs Iohexol Injection in URS
Brief Title: Room Air a Safe Alternative to Dye Injection in Ureterography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, teaching assistant of urology & andrology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: delination of PCS by air
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Ureteral Obstruction
MeSH Terms: conditions — Ureteral Obstruction | interventions — Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with obstructed ureters (Experimental)
  Interventions: Diagnostic Test: air injection

INTERVENTIONS:
Diagnostic Test: air injection — delination of the ureter and pelvis by injecting air under C-ARM

SUMMARY:
The procedure began in the Thirties .Retrograde pyelography is an essential step in most endoscopic procedure. This procedure is used as an investigation, with different indication in the past and the present, to delineate the ureter and pelvicalyceal system either before or after the operation, for example to detect any complication as a perforation and the need for stent placement. The procedure has an alternative, less invasive, the IVP. Multiple articles explored the use of air in the puncture of PCNL and to identify the posterior calyx, but to our knowledge there is no articles addressed the idea of air injection in the ureter. The greatest fear is air embolism or non-visualization of the ureter. The availability and cost of contrast material may be a problem, most urologist face

DETAILED DESCRIPTION:
Our aim is to explore the feasibility of using Room air as a contrast material and check the safety of this procedure.

Materials and methods:

A pilot study in Assiut university hospital Urology department to evaluate the efficacy of air injection as a replacement dye injection in cases of endoscopy either in emergency or elective situation. Twenty patients were selected randomly, to evaluate the impact of retrograde pyelography (RPG) using air in cases of obstructed ureters and raised renal function.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing Urs

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-29 (Estimated); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
no air embolism | 3 months

SECONDARY OUTCOMES:
identification of ureter | intraoperative

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta P, Choudhary GR, Pandey H, Madduri VKS, Singh M, Pallagani L. Air vs contrast pyelogram for initial puncture access in percutaneous nephrolithotomy: a randomized controlled trial. Urolithiasis. 2021 Jun;49(3):261-267. doi: 10.1007/s00240-020-01222-6. Epub 2020 Nov 7. PMID 33159536
- [Background] Sharma AK, Sharma S, Swain S, Goel G, Gujela A, Hota D, Mohapatra B, Sharma B. A comparative study of air pyelogram and contrast pyelogram for initial puncture access and to see its efficacy during percutaneous nephrolithotomy. Urol Ann. 2022 Oct-Dec;14(4):340-344. doi: 10.4103/ua.ua_80_21. Epub 2022 Sep 7. PMID 36505991
- [Background] Jangid DK, Sharma G, Yadav SS, Tomar V, Mathur R. A Comparative Study of Antegrade Air Pyelogram and Retrograde Air Pyelogram for Initial Puncture Access during Percutaneous Nephrolithotomy. J Clin Diagn Res. 2017 Apr;11(4):PC01-PC03. doi: 10.7860/JCDR/2017/24821.9724. Epub 2017 Apr 1. PMID 28571203
- [Background] Garg A, Ali Khan MM, Singh P, Agarwal MK. Air embolism during percutaneous nephrolithotomy using air pyelogram during initial access: Does it really occur? Urol Ann. 2020 Jan-Mar;12(1):54-56. doi: 10.4103/UA.UA_10_19. Epub 2019 Nov 7. PMID 32015618
- [Background] Lipkin ME, Mancini JG, Zilberman DE, Raymundo ME, Yong D, Ferrandino MN, Miller MJ, Yoshizumi TT, Preminger GM. Reduced radiation exposure with the use of an air retrograde pyelogram during fluoroscopic access for percutaneous nephrolithotomy. J Endourol. 2011 Apr;25(4):563-7. doi: 10.1089/end.2010.0431. Epub 2011 Mar 22. PMID 21426236